CLINICAL TRIAL: NCT01329822
Title: The Effects of Caloric Restriction on Fetuin-A and Cardiovascular Risk Factors in Rats and Humans: A Randomized Controlled Trial
Brief Title: Effects of Caloric Restriction on Fetuin-A and Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: Eulji University Hospital (Other)
Responsible Party: Kyung Wan Min, Eulji University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-201104
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes; Overweight
Keywords: type 2 diabetes; overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caloric restriction group (Experimental): CR group were educated by a dietitian to reduce their usual energy intake to 1400 kcal/day (-500 kcal/day, -26% from baseline) for weight reduction and the recommended macronutrient composition was the 50-55% of energy intake as carbohydrate, 15-20% as protein and 20-25% as fat. Daily energy intake and nutrient composition were determined using a computer-aided nutritional analysis program (CAN-Pro 3.0; Korean Nutrition Society, Seoul, South Korea).
  Interventions: Behavioral: Caloric restriction
- Control group (No Intervention): Control group - ad libitum diet

INTERVENTIONS:
Behavioral: Caloric restriction — Caloric restriction
  Arms: Caloric restriction group

SUMMARY:
The aim of this randomized controlled study was to evaluate the effects of CR on circulating fetuin-A levels in obese humans with type 2 diabetes based on monitoring energy intake and energy expenditure by daily activity. Furthermore, the investigators examined the relationship between the changes of fetuin-A levels induced by CR and cardiovascular risk parameters including atherogenic lipid profile, visceral fat area (VFA), brachial artery endothelial function, and carotid IMT.

DETAILED DESCRIPTION:
Rapidly growing aging society augmented the risk of age-associated disorders, such as metabolic syndrome, type 2 diabetes, and cardiovascular disease. Dietary interventions that reduce daily energy intake, also known as caloric restriction (CR), has been shown to be the most robust intervention to extend average and maximal lifespan in various experimental animals (1). In addition, CR diminishes the risk of multiple age-associated diseases, such as diabetes, cardiovascular disease, and some forms of cancer in rodents and primates (rhesus monkeys) (1; 2). Moreover, in obese humans, CR improves insulin sensitivity and reduces fasting glucose as well as the other components of metabolic syndrome (3). However, the exact underlying mechanism of CR has not been fully defined yet.

Recently, it is hypothesized that liver may regulate systemic energy metabolism through production of secretory proteins known as hepatokines. Fetuin-A, a circulating glycoprotein almost exclusively secreted by the liver, has been found to inhibit insulin receptor tyrosine kinase activity in animal studies (4). Fetuin-A knockout (KO) mice have enhanced glucose sensitivity, resistance to weight gain, and lower serum free fatty acid levels (5). In humans, high fetuin-A levels are associated with insulin resistance and fat accumulation in the liver (6). Ix et al. reported that higher human fetuin-A concentrations are strongly associated with metabolic syndrome and atherogenic lipid profile in non-diabetic patients with coronary artery disease (7). In addition, fetuin-A levels were associated with surrogate marker of atherosclerosis such as arterial stiffness and intima-media thickness (IMT) (8). Recent studies reported that elevated fetuin-A levels predict increased risk of myocardial infarction and ischemic stroke (9) as well as type 2 diabetes (10). However, there has been no previous report about the effects of CR on fetuin-A comparing with changes of cardiovascular risk indicators in animals or humans.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI >= 23 kg/m2
* stable body weight (<2 kg change in weight in the past 6 months)
* sedentary lifestyle (<20 min of exercise twice a week)

Exclusion Criteria:

* smoking
* cardiovascular disease
* chronic kidney disease
* chronic liver disease
* pregnant or breast feeding
* any major illness
* taking medications that could affect laboratory test results

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Fetuin-A | 12 weeks
  changes of fetuin-A levels induced by CR

SECONDARY OUTCOMES:
cardiovascular risk factors | 12 weeks
  atherogenic lipid profile, visceral fat area (VFA), brachial artery endothelial function, and carotid IMT.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Wan Min, Principal Investigator — Eulji University
Locations (1):
- Eulji University Hospital, Seoul, South Korea